CLINICAL TRIAL: NCT05952713
Title: Comparative Responses to 15 Different Antidepressants in Major Depressive Disorder - Results From a Long-term Nation-wide Population-based Study Emulating a Randomized Trial
Brief Title: Comparative Responses to 15 Different Antidepressants in Major Depressive Disorder
Status: Completed | Type: Observational
Sponsor: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Sponsor
Other Study IDs: MHSCRDenmark_2
Record Dates: First submitted 2023-07-11; First posted 2023-07-19 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-07

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Antidepressive Agents; Sertraline; Citalopram; Fluoxetine; Paroxetine; Escitalopram; Reboxetine; Venlafaxine Hydrochloride; Duloxetine Hydrochloride; Mirtazapine; Vortioxetine; agomelatine; Amitriptyline; Imipramine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- SSRI: Group 1: Selective serotonin reuptake inhibitors (reference: sertraline)
  Comparisons of the following with sertraline:
  Citalopram, Fluoxetine, Paroxetine, Escitalopram
  Interventions: Drug: Antidepressant
- NARI: Group 2: Noradrenaline reuptake inhibitors (reference: sertraline) Comparisons of the following with sertraline: Reboxetine
  Interventions: Drug: Antidepressant
- SNRI: Group 3: Serotonin and noradrenaline reuptake inhibitors (reference: venlafaxine) Comparisons of Duloxetine with venlafaxine
  Interventions: Drug: Antidepressant
- ARI: Group 4: Adrenergic receptor inhibitors (reference: Mirtazapine) Comparisons of Mianserin with Mirtazapine
  Interventions: Drug: Antidepressant
- Other drugs: Group 5: Other drugs (reference: sertraline) Comparisons of Vortioxetine and Agomelatine with sertraline
  Interventions: Drug: Antidepressant
- TCA: Group 6: Tricyclic antidepressants (reference: amitriptyline)
  Comparisons of Nortriptyline, Imipramine, Clomipramine and Dosulepin with amitriptyline
  Interventions: Drug: Antidepressant

INTERVENTIONS:
Drug: Antidepressant — Treatment with an antidepressant according to Danish register data.
  Other Names: sertraline, citalopram, fluoxetine, paroxetine, escitalopram, reboxetine, venlafaxine, duloxetine, mirtazapine, vortioxetine, agomelatine, amitriptyline, imipramine

SUMMARY:
Achieving results from RCTs with high internal and external validity is a major challenge within psychiatry due to the nature of psychiatric illnesses. The Investigators will conduct a "real world" naturalistic nation-wide population-based longitudinal register linkage study comparing long-term responses to all kinds of antidepressants in patients with major depressive disorder emulating a randomized trial.

ELIGIBILITY:
Inclusion Criteria:

All patients with a psychiatric contact (as inpatients or outpatients) in the period from 1995 to 2018 with a first main index diagnosis of a single depressive episode or recurrent depressive disorder (ICD-10 code: F32-F33.9) with an outpatient purchase of an antidepressant after the depression diagnosis (N=73.336).

Exclusion Criteria:

None.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a psychiatric contact (as inpatients or outpatients) in the period from 1995 to 2018 with a first main index diagnosis of a single depressive episode or recurrent depressive disorder (ICD-10 code: F32-F33.9) with an outpatient purchase of an antidepressant after the depression diagnosis (N=73.336).
Sampling Method: Non-Probability Sample
Enrollment: 73336 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Response | 2 years
  Response was defined as continuous monotherapy with an antidepressant drug without switch to or add-on of another antidepressant drug, an antipsychotic drug or lithium or hospitalization with a main ICD-10 diagnosis of a single depressive episode or recurrent depressive disorder .

CONTACTS AND LOCATIONS:
Locations (1):
- Psychiatric Center Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No